CLINICAL TRIAL: NCT02677311
Title: Gonadotropin Releasing Hormone Agonist (GnRHa) Therapy and Ovarian Preservation in Pediatric and Adolescent Subject Receiving Chemoradiation Therap
Brief Title: GnRHA Therapy and Ovarian Preservation in Pediatric Cancer Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit required numbers for study.
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-0596-F2L
Record Dates: First submitted 2015-12-20; First posted 2016-02-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-05

CONDITIONS: Cancer; Chemoradiation
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Other): Participants who will receive gonadotoxic chemoradiation therapies to include the alkylating agents, heavy metals and plant alkaloids as a standard part of their cancer treatment. Participants will also receive the GnRHa for menstrual suppression as part of standard of care. Baseline blood draws and pelvic ultrasound will be the intervention. Repeat blood draws and pelvic ultrasound at 6 and 12 months will also be interventions.
  Interventions: Procedure: Blood draw; Procedure: Pelvic Ultrasound
- Controls (Other): Participants who will receive chemoradiation therapies presumed to be low risk for gonadotoxicity as determined by the literature and the patient's oncolologist as a standard part of their cancer treatment. Participants will also receive the GnRHa for menstrual suppression as part of standard of care. Baseline blood draws and pelvic ultrasound will be the intervention. Repeat blood draws and pelvic ultrasound at 6 and 12 months will also be interventions.
  Interventions: Procedure: Blood draw; Procedure: Pelvic Ultrasound

INTERVENTIONS:
Procedure: Blood draw — Blood draws will be performed immediately prior to GnRHa treatment and at 6 and 12 months following treatment completion
Procedure: Pelvic Ultrasound — Pelvic ultrasound will be performed immediately prior to GnRHa treatment and at 6 and 12 months following treatment completion

SUMMARY:
This is a prospective case control study. Participants will be enrolled as case subjects or control subjects, depending upon the gonadotoxicity of their chemoradiation therapy. The chemotherapeutic regimens will be determined per standard of care. Participants will receive GnRHa (Lupron) as standard of care for menstrual suppression. Blood draws and pelvic ultrasound at baseline, 6 months and 12 months post completion of chemotherapy are the interventions. The duration of the study will be approximately 12 months.The study time includes the time necessary for completion of most cancer treatments in this population, which approximates 8-12 months, and time to allow complete excretion of the Lupron from the systemic circulation with reliable testing of the hypothalamic pituitary ovarian (H-P-O) axis. The results of the study will be used to guide a larger study evaluating the efficacy of gonadotropin releasing hormone agonist (GnRHa) as ovarian preservation therapy in young subjects receiving chemoradiation.

DETAILED DESCRIPTION:
This study will not utilize a survey or questionnaire. Data will be collected via chart review and direct subject and/or guardian interviews.

Electronic medical records will be accessed only by approved clinical and research personnel to retrieve clinical and laboratory data.

At the initial visit, the following will be performed and collected on all subjects: Body Mass Index; age at thelarche; age at menarche; Tanner staging for breast and pubic hair; oncologic diagnosis; date of oncologic diagnosis; chemoradiation therapy treatment regimen; date of initiation of chemoradiation therapy; pre-treatment ovarian function blood tests; date GnRHa therapy initiated; a pelvic ultrasound will be performed to assess ovarian volumes and antral follicle count.

The subject will receive GnRHa 11.25 mg every 2 months until completion of chemotherapy, which is consistent with current clinical care at the University of Kentucky Medical Center (UKMC).

Study blood tests to evaluate ovarian function and pelvic ultrasound will be performed at three time points: immediately prior to initiation of GnRHa therapy and 6 and 12 months after chemoradiation therapy is completed.

The subject/guardian will be contacted by the study team at regular intervals to assess her progress and plan timing of study visits.

At subsequent visits, the investigator will record the date chemoradiation therapy treatment ended; date and reason GnRHa therapy discontinued; presence of breakthrough bleeding (BTB); timing of BTB in relation to most recent GnRHa injection. In order to document bleeding patterns, subjects will be asked to fill out the pictorial assessment of bleeding chart every month that they are in the study.

Six months after completion of chemoradiation therapy, the investigator will assess post-treatment ovarian function blood test levels and performed a pelvic U/S to assess ovarian volumes and antral follicle count. Investigator will as assess the resumption of spontaneous menses, parity, date of subject demise, if applicable.

Twelve months after completion of chemotherapy, we will assess post-treatment ovarian function blood test levels; and performed a pelvic U/S to assess ovarian volumes and antral follicle count. Investigator will as assess the resumption of spontaneous menses, parity, date of subject demise, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemoradiation therapy
* Documented ovarian function
* Require menstrual suppression with GnRHa during chemoradiation therapy
* Patients at the University of Kentucky, Norton Healthcare or Cincinnati Children's Hospital Medical Center

Exclusion Criteria:

* Under 8 years of age and older than 19 years of age
* Male
* Unable to provide consent or assent

Ages: 8 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Ovarian Reserve - AMH | 6 months post completion of chemotherapy
  Assess AMH change from baseline to 6 months.
Ovarian Reserve - AMH | 12 months post completion of chemotherapy
  Assess AMH change from baseline to 12 months.
Ovarian Reserve - Menstrual function | 12 months post completion of chemotherapy
  Assess menstrual function change from baseline to 12 year.
Ovarian Reserve - FSH | 6 months post completion of chemotherapy
  Assess FSH change from baseline to 6 months.
Ovarian Reserve - FSH | 12 months post completion of chemotherapy
  Assess FSH change from baseline to 12 months.
Ovarian Reserve - Menstrual function | 6 months post completion of chemotherapy
  Assess menstrual function change from baseline to 6 months.

SECONDARY OUTCOMES:
Ovarian Reserve - Agreement of AMH and AFC | Pre-GnRHa therapy, 6 months post and 12 post completion of chemotherapy
  To assess the agreement of AMH (< or equal to 0.5 vs. > 0.5) and AFC (<16 follicles vs 16+ follicles) as indicators of ovarian reserve after chemoradiation and GnRHa therapy

IPD SHARING:
Plan to Share IPD: Yes
* UK IRB/Office of Research Integrity
  * Law enforcement agencies when required by law
  * University of Kentucky representatives
  * UK Hospital
  * ACOG
  * Representatives of the National Cancer Institute (NCI), FDA, and other U.S. and international governmental regulatory agencies involved in overseeing research
  * Authorized representatives at the University of Cincinnati who are collaborating on this research.
  * Every research site of the study (including UK Healthcare and Cincinnati Children's and each site's research staff and medical staff)
  * Every health care provider who provides services to you in connection with the study
  * Any laboratories and other individuals and organizations that analyze your PHI in connection with the study
  * The Sponsor and the people and companies they use to oversee, administer and/or conduct the study
  * Kentucky Cancer Registry (KCR) to all follow-up assistance